CLINICAL TRIAL: NCT02674555
Title: A Phase 1 Study to Investigate the Absorption, Metabolism and Excretion of [14C]ASP8273 in Subjects With Solid Tumors Harboring Epidermal Growth Factor Receptor (EGFR) Mutations
Brief Title: A Study to Investigate the Absorption, Metabolism and Excretion of [14C]ASP8273 in Subjects With Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Following recommendation by SOLAR Study IDMC, Astellas closed enrollment in ASP8273 studies.
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8273-CL-0104
Record Dates: First submitted 2016-01-21; First posted 2016-02-04 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Epidermal Growth Factor Receptor (EGFR) Mutations; Solid Tumors
Keywords: Phase 1; Metabolism; Excretion; Absorption; [14C]-radioactivity; Pharmacokinetics; naquotinib; Oncology
MeSH Terms: conditions — Neoplasms | interventions — naquotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP8273 (Experimental): Two Parts - Part A: 14C-radio labeled; Part B: non radio labeled (optional)
  Interventions: Drug: radio-labeled naquotinib; Drug: naquotinib

INTERVENTIONS:
Drug: radio-labeled naquotinib — Oral administration
  Other Names: ASP8273
Drug: naquotinib — Oral administration
  Other Names: ASP8273

SUMMARY:
This is a study to investigate the absorption, metabolism and excretion of [14C] labeled ASP8273 in subjects with solid tumors harboring EGFR mutations (per local testing). This study consists of two parts (A and B).

DETAILED DESCRIPTION:
This study consists of two parts (A and B).

In Part A, eligible subjects will be admitted to the site on day -1 and remain confined at the site until postdosing discharge criteria are met. Subjects will receive a single dose of [14C] ASP8273 solution on study day 1.

Once Part A has been completed, subjects may elect to continue participation in Part B. Subjects will receive oral administration of ASP8273 (nonradiolabeled) once daily in 28-day cycles.

ELIGIBILITY:
Inclusion Criteria:

* Subject has histologically or cytologically confirmed metastatic or locally advanced, unresectable solid tumors harboring EGFR mutations.
* Subject has Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
* Subject must meet all of the following criteria on the laboratory tests that will be performed within 7 days prior to enrollment. In case of multiple laboratory data within this period, the most recent data should be used.

  * Neutrophil count ≥ 1,000/mm3
  * Platelet count ≥ 7.5 × 104/mm3
  * Hemoglobin ≥ 9.0 g/dL
  * Lymphocyte count ≥ 500/mm3
  * Estimated glomerular filtration rate (eGFR) of > 50 ml/min as calculated by the Cockcroft-Gault Method
  * Total bilirubin (TBL) < 1.5 × upper limit of normal (ULN; except for subjects with documented Gilbert's syndrome)
  * Aspartate aminotransferase (AST) and ALT < 3.0 × ULN
  * Serum sodium level is ≥ 130 mmol/L
* Female subject must either be:

  * Of nonchild bearing potential:

    1. Postmenopausal (defined as at least 1 year without any menses) prior to screening, or
    2. Documented surgically sterile or status post hysterectomy (at least 1 month prior to screening).
  * Or, if of childbearing potential:

    1. Agree not to try to become pregnant during the study and for 28 days after the final study drug administration,
    2. Must have a negative serum pregnancy test at screening and day -1, and
    3. If heterosexually active must use two forms of birth control* (at least one of which must be a barrier method) starting at screening and throughout the study period and for 28 days after the final study drug administration.
* Female subject must not be breastfeeding at screening or during the study period, and for 28 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 28 days after the final study drug administration.
* Male subject and his female spouse/partner who is of childbearing potential must be using highly effective contraception consisting of two forms of birth control* (one of which must be a barrier method) starting at screening and continue throughout the study period and for 90 days after the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period and for 90 days after the final study drug administration.

  *Acceptable forms of birth control include:
* Established use of oral, injected or implanted hormonal methods of contraception.
* Placement of an intrauterine device (IUD) or intrauterine system (IUS).
* Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.

Exclusion Criteria:

* Subject has an ongoing toxicity ≥ Grade 2 (Common Terminology Criteria for Adverse Event [CTCAE] v4.03) attributable to prior medication to treat solid tumor (except alopecia) at the time of screening.
* Subject has known history of serious hypersensitivity reaction to ASP8273, or any component of the formulation used.
* Subject has received investigational therapy within 28 days or 5 half-lives, whichever is shorter, prior to the first dose of study drug.
* Subject has received a prior EGFR inhibitor within 6 days prior to the first dose of study drug.
* Subject has had any of the following within 14 days prior to the first dose of study drug:

  * A treatment with any other agent with antitumor activity including chemotherapy, radiotherapy, or immunotherapy
  * A major surgical procedure (other than study related biopsy), or a major surgical is planned to occur during the study
  * Blood transfusions or hemopoietic factor therapy
  * Evidence of active infection requiring systemic therapy
* Subject has symptomatic central nervous system (CNS) metastasis. Subject with previously treated brain or CNS metastases are eligible provided that the subject has recovered from any acute effects of radiotherapy and is not requiring steroids, and any whole brain radiation therapy was completed at least 2 weeks prior to study drug administration, or any stereotactic radiosurgery (SRS) was completed at least 1 week prior the first dose of study drug.
* Subject has ≥ CTCAE v4.03 Grade 2 neuropathy.
* Subject has a known history of a positive test for hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV).
* Subject has a known history of a positive test for human immunodeficiency virus (HIV) infection.
* Subject has history of drug-induced interstitial lung disease (ILD) or any evidence of active ILD.
* Subject has severe or uncontrolled systemic diseases including uncontrolled hypertension (blood pressure > 150/100 mmHg) or active bleeding diatheses.
* Subject has ongoing cardiac arrhythmia that is Grade ≥ 2 or uncontrolled atrial fibrillation of any grade.
* Subject currently has Class 3 or 4 New York Heart Association congestive heart failure.
* Subject has history of severe/unstable angina, myocardial infarction, or cerebrovascular accident within 6 months prior to the first dose of study drug.
* Subject has concurrent corneal disorder or any ophthalmologic condition which, in the Investigator's opinion, makes the subject unsuitable for study participation (e.g., advanced cataracts, glaucoma, or subject is unable to undergo a comprehensive ophthalmologic exam).
* Subject has history of gastrointestinal ulcer or gastrointestinal bleeding within 3 months prior to the first dose of study drug.
* Subject has difficulty taking oral medication or any digestive tract dysfunction or inflammatory bowel disease that would interfere with the intestinal absorption of drug.
* Subject who has received strong/moderate inhibitors or inducers of CYP3A4 within 14 days prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-15 (Actual)

PRIMARY OUTCOMES:
Part A: Radioactivity in whole blood: AUCinf | Up to 14 days
  AUCinf: area under the concentration-time curve from the time of dosing extrapolated to time infinity
Part A: Radioactivity in whole blood: AUClast | Up to 14 days
  AUClast: area under the concentration-time curve from the time of dosing to the last measurable concentration
Part A: Radioactivity in whole blood: Cmax | Up to 14 days
  Cmax: maximum concentration
Part A: Radioactivity in whole blood: tmax | Up to 14 days
  tmax: time to maximum concentration
Part A: Radioactivity in whole blood: t1/2 | Up to 14 days
  t1/2: apparent terminal elimination half-life
Part A: Radioactivity in plasma: AUCinf | Up to 14 days
Part A: Radioactivity in plasma: AUClast | Up to 14 days
Part A: Radioactivity in plasma: Cmax | Up to 14 days
Part A: Radioactivity in plasma: tmax | Up to 14 days
Part A: Radioactivity in plasma: t1/2 | Up to 14 days
Part A: Radioactivity ratio for whole blood/plasma concentration (per time point.) | Up to 14 days
Part A: Radioactivity ratio for whole blood/plasma AUCinf | Up to 14 days
Part A: Radioactivity ratio for whole blood/plasma AUClast | Up to 14 days
Part A: Excretion ratio of radioactivity in urine | Up to 14 days
Part A: Cumulative excretion of radioactivity in urine | Up to 14 days
Part A: Excretion ratio of radioactivity in feces | Up to 14 days
Part A: Cumulative excretion of radioactivity in feces | Up to 14 days
Part A: Total excretion ratio of radioactivity in urine and feces | Up to 14 days
Part A: Total cumulative excretion of radioactivity in urine and feces | Up to 14 days
Part A: Radioactivity in emesis (if applicable) | Up to 14 days
Part A: Pharmacokinetics of ASP8273 and possible metabolites in plasma: AUCinf | Up to 14 days
Part A: Pharmacokinetics of ASP8273 and possible metabolites in plasma: AUClast | Up to 14 days
Part A: Pharmacokinetics of ASP8273 and possible metabolites in plasma: Cmax | Up to 14 days
Part A: Pharmacokinetics of ASP8273 and possible metabolites in plasma: tmax | Up to 14 days
Part A: Pharmacokinetics of ASP8273 and possible metabolites in plasma: t1/2 | Up to 14 days
Part A: Pharmacokinetics of ASP8273 and possible metabolites in urine: (Aelast) | Up to 14 days
  Aelast: cumulative amount of drug excreted from time of dosing up to the collection time of the last measurable concentration
Part A: Pharmacokinetics of ASP8273 and possible metabolites in urine CLr | Up to 14 days
  CLr: renal clearance
Part A: Pharmacokinetics of ASP8273 and possible metabolites in urine: % of dose excreted (Aelast%) | Up to 14 days

SECONDARY OUTCOMES:
Part A: Profiling of possible metabolites of ASP8273 in plasma | Up to 14 days
  Identification and possible quantification of metabolites in plasma
Part A: Profiling of possible metabolites of ASP8273 in urine | Up to 14 days
  Identification and possible quantification of metabolites in urine
Part A: Profiling of possible metabolites of ASP8273 in feces | Up to 14 days
  Identification and possible quantification of metabolites in feces
Part A and Part B: Safety profile assessed by adverse event reporting, vital signs, electrocardiograms (ECG), clinical laboratory tests, and physical examinations | Up to 36 months
  Vital signs include oral temperature, pulse, and blood pressure. Clinical laboratory evaluations include hematology, chemistry and urinalysis.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.

IPD SHARING:
Plan to Share IPD: Undecided